CLINICAL TRIAL: NCT00059202
Title: Multicentered Randomized Trial of High-dose Urso in Primary Sclerosing Cholangitis
Brief Title: Trial of High-dose Urso in Primary Sclerosing Cholangitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: DSMB reviewed interim analysis and terminated the study due to futility.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: URSO (completed); R01DK056924 (NIH)
Record Dates: First submitted 2003-04-21; First posted 2003-04-22 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Urso; PSC
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet that is identical (size, color, etc) to experimental ursodeoxycholic acid tablet.
  Interventions: Drug: Placebo
- Ursodeoxycholic acid (Experimental): Ursodeoxycholic acid 28-30 mg/kg/day
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Ursodeoxycholic Acid 28-30 mg/kg/day in divided doses
  Other Names: UDCA
  Arms: Ursodeoxycholic acid
Drug: Placebo — Placebo for Urso
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, controlled trial of high dose ursodiol versus placebo for patients with primary sclerosing cholangitis (PSC). The average duration of follow-up will be approximately five years with important clinical endpoints such as death, eligibility for liver transplantation, changes in histology and cholangiogram as well as liver biochemistries and quality of life data collected.

ELIGIBILITY:
* Chronic cholestatic disease of at least six months' duration.
* Serum alkaline phosphatase at least 1 ½ times the upper limits of normal.
* Retrograde, operative, percutaneous, or magnetic resonance cholangiography demonstrating intrahepatic and/or extrahepatic biliary duct obstruction, beading, or narrowing consistent with PSC within one year of the study entry.
* Liver biopsy in the previous one year which is available for review and compatible with the diagnosis of PSC. Compatible biopsy features include fibrous cholangitis, ductopenia with periportal inflammation and biliary fibrosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Medical College of Virginia, Richmond, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Lindor KD, Kowdley KV, Luketic VA, Harrison ME, McCashland T, Befeler AS, Harnois D, Jorgensen R, Petz J, Keach J, Mooney J, Sargeant C, Braaten J, Bernard T, King D, Miceli E, Schmoll J, Hoskin T, Thapa P, Enders F. High-dose ursodeoxycholic acid for the treatment of primary sclerosing cholangitis. Hepatology. 2009 Sep;50(3):808-14. doi: 10.1002/hep.23082. PMID 19585548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ursodeoxycholic Acid | Placebo
Started | 76 | 74
Completed | 70 | 59
Not Completed | 6 | 15
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Protocol Violation | 1 | 3
Not completed — drug toxicity | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ursodeoxycholic Acid | Placebo | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Continuous [Median (Full Range); unit: years] | 47.9 [20.5 to 75.6] | 45.3 [17.9 to 73.6] | 46.6 [17.9 to 75.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 26 | 64
  Male | 38 | 48 | 86
Region of Enrollment [Number; unit: participants]
  United States | 76 | 74 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure was defined as death, transplantation, meeting minimal listing criteria, development of varices, cholangiocarcinoma, or progression to cirrhosis
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 76 | 74
Participants | 30 | 19

2. Secondary Outcome: Number of Deaths
Description: Death at any time up to 5 years
Time Frame: 5 years
Measure: Number; unit: participants
Groups:
- Placebo: Placebo or Urso
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 76 | 74
participants | 5 | 3

3. Secondary Outcome: Number of Participants Who Have a Liver Transplantation
Description: Liver transplantation at any time up to 5 years
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 76 | 74
participants | 11 | 5

4. Secondary Outcome: Number of Participants Meeting Minimal Listing Criteria for Liver Transplantation
Description: Meeting minimal listing criteria for liver transplantation at any time up to 5 years. Minimal listing criteria are defined as a MELD score of 14 or higher. The Model For End-Stage Liver Disease (MELD) is a numeric score with a range of 6 to 40, where a higher score means worse liver disease.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 76 | 74
participants | 13 | 10

5. Secondary Outcome: Number of Participants Who Developed Cholangiocarcinoma
Description: Development of cholangiocarcinoma at any time up to 5 years
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 76 | 74
participants | 2 | 2

6. Secondary Outcome: Number of Participants Who Developed Varices
Description: Development of esophogeal and/or gastric varices
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 76 | 74
participants | 15 | 5

7. Secondary Outcome: Number of Participants Who Developed Cirrhosis
Description: Development of cirrhosis based on liver biopsy
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 76 | 74
participants | 6 | 4

8. Secondary Outcome: Alkaline Phosphatase at 12 Months
Description: Alkaline phosphatase divided by the upper limit of normal
Time Frame: 12 months
Measure: Median (Full Range); unit: Ratio
Groups:
- Placebo: Identical placebo
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 70 | 63
Ratio | 1.9 [0.6 to 9.1] | 2.9 [0.6 to 13.6]

9. Secondary Outcome: Alkaline Phosphatase at 24 Months
Description: Alkaline phosphatase divided by the upper limit of normal
Time Frame: 24 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 65 | 58
Ratio | 1.8 [0.6 to 8.5] | 2.6 [0.5 to 11.9]

10. Secondary Outcome: Alkaline Phosphatase at 36 Months
Description: Alkaline phosphatase divided by the upper limit of normal
Time Frame: 36 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 56 | 53
Ratio | 1.7 [0.6 to 16.5] | 2.4 [0.4 to 12.1]

11. Secondary Outcome: Aspartate Aminotransferase at 12 Months
Description: Aspartate aminotransferase at divided by the upper limit of normal
Time Frame: 12 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 70 | 63
Ratio | 1.0 [0.5 to 10.5] | 1.9 [0.6 to 8.7]

12. Secondary Outcome: Aspartate Aminotransferase at 24 Months
Description: Aspartate aminotransferase at divided by the upper limit of normal
Time Frame: 24 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 65 | 59
Ratio | 1.1 [0.4 to 8.4] | 1.9 [0.5 to 13.3]

13. Secondary Outcome: Aspartate Aminotransferase at 36 Months
Description: Aspartate aminotransferase at divided by the upper limit of normal
Time Frame: 36 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 56 | 53
Ratio | 1.1 [0.3 to 7.2] | 1.7 [0.5 to 14.8]

14. Secondary Outcome: Bilirubin at 12 Months
Description: Bilirubin divided by the upper limit of normal
Time Frame: 12 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 70 | 63
Ratio | 0.8 [0.2 to 6.3] | 0.9 [0.3 to 8.2]

15. Secondary Outcome: Bilirubin at 24 Months
Description: Bilirubin divided by the upper limit of normal
Time Frame: 24 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 64 | 59
Ratio | 0.8 [0.2 to 7.2] | 1.0 [0.2 to 8.6]

16. Secondary Outcome: Bilirubin at 36 Months
Description: Bilirubin divided by the upper limit of normal
Time Frame: 36 months
Measure: Median (Full Range); unit: Ratio
Arm/Group | Ursodeoxycholic Acid | Placebo
Number analyzed (Participants) | 55 | 53
Ratio | 0.8 [0.2 to 15.9] | 0.9 [0.3 to 9.6]

ADVERSE EVENTS:
Time Frame: Five years
Arm/Group | Ursodeoxycholic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 5/76 | 3/74
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No